CLINICAL TRIAL: NCT03866473
Title: A Pilot Study Evaluating Photobiomodulation Therapy for Diabetic Macular Edema
Acronym: AE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Eye Institute (NEI) (NIH); Juvenile Diabetes Research Foundation (Other); PhotoOptx LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRCR.net Protocol AE
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Results first posted 2022-06-10 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Random assignment (1:1) to photobiomodulation (PBM) or sham
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Optical coherence tomography technicians and visual acuity testers, including refractionists, will be masked to treatment group at outcome visits. Study participants will be masked to their treatment group assignment. Every effort will be made to keep investigators masked. Study coordinators who will be involved with training and compliance assessment will not be masked to treatment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Photobiomodulation (PBM) (Experimental): 670nm wavelength device twice a day for 90 seconds through 4 months. At the 4-month visit, participants who have not already received alternative treatments for DME will return the original device and receive the alternative treatment group device (i.e. the sham group will receive an active treatment device and the active treatment group will receive a sham device).
  Interventions: Device: Retilux
- Placebo (Sham Comparator): Broad spectrum light device twice a day for 90 seconds through 4 months. At the 4-month visit, participants who have not already received alternative treatments for DME will return the original device and receive the alternative treatment group device (i.e. the sham group will receive an active treatment device and the active treatment group will receive a sham device)
  Interventions: Device: Sham Light Device

INTERVENTIONS:
Device: Retilux — 670nm wavelength light
  Other Names: PBM; Photobiomodulation
  Arms: Photobiomodulation (PBM)
Device: Sham Light Device — Broad spectrum light device
  Arms: Placebo

SUMMARY:
Randomized clinical trial evaluating the effect of photobiomodulation compared with sham on central subfield thickness (CST) in eyes with central-involved DME and good vision.

DETAILED DESCRIPTION:
This study is being conducted to assess the effects of photobiomodulation on CST compared with sham in eyes with central-involved DME and good vision. Photobiomodulation is irradiation by light in the 630-900 nanometer region of the spectrum.

Furthermore, this pilot study is being conducted to determine whether the conduct of a pivotal trial has merit based on an anatomic outcome and provide information on outcome measures needed to design a pivotal trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of diabetes mellitus (type 1 or type 2). Any one of the following will be considered to be sufficient evidence that diabetes is present:

  1. Current regular use of insulin for the treatment of diabetes.
  2. Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes.
  3. Documented diabetes by American Diabetes Association and/or the World Health Organization criteria.
  4. Able and willing to provide informed consent.

Atleast one eye meeting the following criteria:

1. Best corrected E-ETDRS visual acuity letter score ≥ 79 (i.e., 20/25 or better)
2. Ophthalmoscopic evidence of central-involved DME, confirmed by CST on spectral domain OCT: Zeiss Cirrus: ≥290µm in women, and ≥305µm in men, Heidelberg Spectralis: ≥305µm in women, and ≥320µm in men
3. Media clarity, pupillary dilation, and study participant

Exclusion Criteria:

* History of chronic renal failure requiring dialysis or kidney transplant.
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status that might preclude completion of follow-up).
* Initiation of intensive insulin treatment (a pump or multiple daily injections) within 4 months prior to randomization or plans to do so in the next 4 months.
* Participation in an investigational trial that involved treatment within 30 days of randomization with any drug/device that has not received regulatory approval for the indication being studied. Note: study participants cannot participant in another investigational trial that involves treatment with an investigational drug or device while participating in the study.
* Systolic blood pressure above 180 or diastolic blood pressure above 110. If blood pressure is brought below 180 systolic and 110 diastolic by anti-hypertensive treatment, individual can become eligible.
* Systemic anti-vascular endothelial growth factor (anti-VEGF) or pro-VEGF treatment within 4 months prior to randomization. These drugs should not be used during the study.
* For women of child-bearing potential: pregnant or intending to become pregnant within the next 8 months. Women who are potential study participants should be questioned about the potential for pregnancy. Investigator judgment is used to determine when a pregnancy test is needed.
* Individual is expecting to move out of the area during the 8 months of the study.

A participant will be excluded if the study eye meets any of the following criteria:

* Macular edema is considered to be due to a cause other than DME. An eye should not be considered eligible if: (1) the macular edema is considered to be related to ocular surgery such as cataract extraction or (2) clinical exam and/or investigator assessment of OCT suggests that vitreoretinal interface abnormalities (e.g., a taut posterior hyaloid or epiretinal membrane) are contributing to the macular edema.
* An ocular condition is present such that, in the opinion of the investigator, any visual acuity loss would not improve from resolution of macular edema (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, nonretinal condition).
* An ocular condition is present (other than DME) that, in the opinion of the investigator, might affect visual acuity during the course of the study or require intraocular treatment (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.)
* Cataract is present that, in the opinion of the investigator, may alter visual acuity during the course of the study.
* History of major ocular surgery (including cataract, scleral buckle, any intraocular surgery, etc.) within prior 4 months or major ocular surgery anticipated during the study period.
* Any history of prior laser or other surgical, intravitreal, or peribulbar treatment for DME or DR (such as panretinal photocoagulation, focal/grid macular photocoagulation, intravitreal or peribulbar corticosteroids, or anti-VEGF) within the prior 12 months. If treatment was given more than 12 months prior, no more than 4 prior intraocular injections. Enrollment will be limited to a maximum of 15 percent of the planned sample size with any history of anti-VEGF treatment and a maximum of 15% with any history of PRP.
* Anticipated need to treat DME or DR during the study period
* History of topical steroid or non-steroidal anti-inflammatory drug treatment within 30 days prior to randomization.
* History of YAG capsulotomy performed within 2 months prior to randomization
* Any history of vitrectomy.
* Aphakia
* Uncontrolled glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy Kim, MD, Study Chair — Medical College of Wisconsin Eye Institute
Locations (20):
- United States (20):
  - Atlantis Eye Care, Huntington Beach, California
  - East Bay Retina Consultants, Inc, Oakland, California
  - California Retina Consultants, Santa Barbara, California
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - UF College of Medicine, Dept of Ophthalmology, Jacksonville Health Science Center, Jacksonville, Florida
  - Southeast Retina Center, PC, Augusta, Georgia
  - Marietta Eye Clinic, Marietta, Georgia
  - Raj K. Maturi, MD, PC, Indianapolis, Indiana
  - Mid-America Retina Consultants, PA, Overland Park, Kansas
  - Paducah Retinal Center, Paducah, Kentucky
  - Elman Retina Group, PA, Baltimore, Maryland
  - Mid Atlantic Retina Specialists, Hagerstown, Maryland
  - Valley Eye Physicians and Surgeons, Ayer, Massachusetts
  - The Retina Institute, St Louis, Missouri
  - Charlotte Eye, Ear, Nose and Throat Assoc., PA, Charlotte, North Carolina
  - Retina Northwest PC, Portland, Oregon
  - Southeastern Retina Associates, PC, Knoxville, Tennessee
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, Austin, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Visit completion at 4 months was prespecified as completion of any study visit from 12 to 24 weeks but due to the COVID19 pandemic, the window was extended to 32 weeks and participants in Phase 2 could also discontinue device use.
Units Other Than Participants: Eyes
Groups:
- Photobiomodulation (PBM) Intervention: 670nm wavelength device twice a day for 90 seconds through 4 months. At the 4-month visit, participants who have not already received alternative treatments for DME will return the original device and receive the alternative treatment group device (i.e. the sham group will receive an active treatment device and the active treatment group will receive a sham device).
  Retilux: 670nm wavelength light
- Placebo Intervention: Broad spectrum light device twice a day for 90 seconds through 4 months. At the 4-month visit, participants who have not already received alternative treatments for DME will return the original device and receive the alternative treatment group device (i.e. the sham group will receive an active treatment device and the active treatment group will receive a sham device)
  Sham Light Device: Broad spectrum light device
Period: Phase 1
Arm/Group | Photobiomodulation (PBM) Intervention | Placebo Intervention
Started | 69; 69 Eyes | 66; 66 Eyes
Completed | 68; 68 Eyes | 66; 66 Eyes
Not Completed | 1; 1 Eyes | 0; 0 Eyes
Not completed — Death | 1 | 0
Period: Phase 2
Arm/Group | Photobiomodulation (PBM) Intervention | Placebo Intervention
Started | 62; 62 Eyes (Three participants completed the study by receiving alternate treatment for diabetic macular edema in phase 1 and 3 were dropped.) | 61; 61 Eyes
Completed | 60; 60 Eyes | 58; 58 Eyes (One participant completed the study by receiving alternate treatment for diabetic macular edema in Phase 1 and 4 participants were dropped.)
Not Completed | 2; 2 Eyes | 3; 3 Eyes
Not completed — Death | 0 | 2
Not completed — Dropped | 1 | 1
Not completed — Completed the study by receiving alternate treatment for diabetic macular edema | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Photobiomodulation (PBM) | Placebo | Total
Number analyzed (Participants) | 69 | 66 | 135
Age, Customized [Median (Inter-Quartile Range); unit: years] | 63 [55 to 66] | 62 [58 to 69] | 62 [56 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 28 | 50
  Male | 47 | 38 | 85
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1
  Black/African American | 4 | 7 | 11
  Hispanic or Latino | 5 | 7 | 12
  White | 59 | 52 | 111
Diabetes Type [Number; unit: participants]
  Type 1 | 5 | 10 | 15
  Type 2 | 64 | 56 | 120
Hemoglobin A1c [Number; unit: participants] — Population: Hemoglobin A1c was missing for 2 PBM and 2 placebo participants.
  participants
    Less than 7.5%: number analyzed (Participants) | 67 | 64 | 131
    Less than 7.5% | 33 | 23 | 56
    7.5% or more: number analyzed (Participants) | 67 | 64 | 131
    7.5% or more | 34 | 41 | 75
E-ETDRS visual acuity letter score [Median (Inter-Quartile Range); unit: units on a scale] — Best-corrected visual acuity following protocol-defined refraction. Visual Acuity was measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/10) to 0 letters (Snellen equivalent <20/800). Higher scores indicate better visual acuity and lower scores indicate worse visual acuity.
  units on a scale | 84.0 [81.0 to 87.0] | 85.0 [82.0 to 88.0] | 84 [81 to 87]
Optical coherence tomography central subfield thickness [Median (Inter-Quartile Range); unit: Microns] — Spectralis equivalent. Cirrus measurements were converted to Spectralis equivalents using the following formula: Spectralis = 40.78 +0.95 x Cirrus
  Microns | 352 [335 to 387] | 355 [337 to 374] | 354 [335 to 378]
Lens Status on Clinical Exam [Number; unit: participants]
  Phakic (natural lens) | 19 | 15 | 34
  Prosthetic intraocular lens | 50 | 51 | 101
Diabetic retinopathy severity [Number; unit: participants] — NPDR= Non-proliferative diabetic retinopathy
  participants
    Microaneurysms only | 0 | 1 | 1
    Mild/moderate NPDR | 58 | 48 | 106
    Severe NPDR | 7 | 11 | 18
    Proliferative diabetic retinopathy or prior scatter laser or both. | 4 | 6 | 10
Atleast one prior treatment for diabetic macular edema [Number; unit: participants] | 15 | 12 | 27
Retinal Volume [Median (Inter-Quartile Range); unit: mm^3] — Measured on optical coherence tomography
  mm^3 | 7.72 [7.19 to 8.15] | 7.68 [7.12 to 8.12] | 7.70 [7.19 to 8.17]
Iris color [Number; unit: Eyes]
  Blue | 19 | 28 | 47
  Brown | 31 | 27 | 58
  Other | 19 | 11 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Optical Coherence Tomography Central Subfield Thickness From Baseline to 4 Months
Description: Only eyes that completed the 4-month visit were included in calculation of descriptive statistics of optical coherence tomography (OCT) data. For eyes that received alternate DME treatment prior to 4 months (N=3 [PBM]; N = 1 [placebo]), the last OCT measurements prior to alternative diabetic macular edema (DME) treatment were used in place of the 4-month measurements. All analyses followed the intent-to-treat principle. Multiple imputation (m = 100) was used for missing values of central subfield thickness and retinal volume change, with imputation models that included variables for treatment group, baseline values, and change from baseline at all monthly interim visits up to the primary outcome visit and the randomization stratification factor of recent or planned intravitreous treatment in the non-study eye. Multiple imputation was not performed for center-involved DME given the thresholds are gender and machine specific.
  OCT CST change was truncated to the mean ± 3 SD (13 ± 3 × 5
Time Frame: Baseline to 4 months
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Arm/Group | Photobiomodulation (PBM) | Placebo
Number analyzed (Participants) | 68 | 66
Number analyzed (Eyes) | 68 | 66
microns | 13 (53) | 15 (57)

2. Secondary Outcome: Mean Change in Retinal Volume on Optical Coherence Tomography From Baseline to 4 Months
Description: CST = central subfield thickness, OCT = optical coherence tomography, PBM = photobiomodulation
Time Frame: Baseline to 4 months
Population: Multiple imputation (m=100) was used for missing values of CST and retinal volume change, with imputation models that were stratified by treatment and included variables for treatment group, baseline values, and change from baseline at all monthly interim visits up to the primary outcome visit and the randomization stratification factor of recent or planned intravitreous treatment in the non-study eye. OCT retinal volume change was missing for 8 PBM and 5 placebo eyes.
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Eyes
Arm/Group | Photobiomodulation (PBM) | Placebo
Number analyzed (Participants) | 60 | 61
Number analyzed (Eyes) | 60 | 61
mm^3 | 0.12 (0.45) | 0.10 (0.42)

3. Secondary Outcome: Number of Eyes With Center-involved Diabetic Macular Edema on Optical Coherence Tomography at 4 Months
Description: DME = diabetic macular edema, OCT = optical coherence tomography
Time Frame: baseline to 4 months
Population: Eyes that received alternate DME treatment (N = 3 (Photobiomodulation); N = 1 (Placebo)) used the last OCT measurement prior to receiving treatment. Missing values were not imputed.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Photobiomodulation (PBM) | Placebo
Number analyzed (Participants) | 68 | 66
Number analyzed (Eyes) | 68 | 66
Eyes | 61 | 57

4. Secondary Outcome: Number of Eyes Receiving Alternative Treatment for Diabetic Macular Edema
Time Frame: 4 months
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Photobiomodulation (PBM) | Placebo
Number analyzed (Participants) | 68 | 66
Number analyzed (Eyes) | 68 | 66
Eyes | 3 | 1

5. Secondary Outcome: Change in Visual Acuity From Baseline to 4 Months
Description: Visual acuity is measured as a continuous integer letter score from 0 to 100, with higher numbers indicating better visual acuity. A letter score of 85 is approximately 20/20 and a letter score of 70 is approximately 20/40, the legal unrestricted driving limit in most states. A 5-letter change for an individual is approximately equal to a 1-line change on a vision chart. Visual acuity (VA) change truncated to mean ±3 SD (-0.3 ± 3 × 5.3). Eyes that received alternative treatment for DME before primary outcome visit (3 PBM, 1 placebo); last measurements taken before DME treatment was initiated were the pre-specified outcome data. Missing data for eyes that didn't get alternative treatment for DME imputed with multiple imputation.
Time Frame: baseline to 4 months
Population: Multiple imputation (m=100) used for missing values of VA change, with imputation models that were stratified by treatment and included variables for baseline VA, change from baseline at all monthly interim visits up to the primary outcome visit and the randomization stratification factor of recent or planned intravitreous treatment in the non-study eye.
Measure: Mean (Standard Deviation); unit: Letter Score
Units Other Than Participants: Eyes
Arm/Group | Photobiomodulation (PBM) | Placebo
Number analyzed (Participants) | 68 | 66
Number analyzed (Eyes) | 68 | 66
Letter Score | -0.2 (5.5) | -0.6 (4.6)

6. Secondary Outcome: Change in Optical Coherence Tomography Central Subfield Thickness From 4 to 8 Months
Description: Only eyes that completed the 4-month visit were included in calculation of descriptive statistics of OCT data. For eyes that received alternate DME treatment prior to 4 months (N = 3 [PBM]; N = 1 [placebo]), the last OCT measurements prior to alternative DME treatment were used in place of the 4-month measurements. All analyses followed the intent-to-treat principle. Multiple imputation (m = 100) was used for missing values of central subfield thickness and retinal volume change, with imputation models that included variables for treatment group, baseline values, and change from baseline at all monthly interim visits up to the primary outcome visit and the randomization stratification factor of recent or planned intravitreous treatment in the non-study eye. Multiple imputation was not performed for center-involved DME given the thresholds are gender and machine specific.
  OCT CST change was truncated to the mean ± 3 SD (13 ± 3 × 58)
Time Frame: 4 to 8 months
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Groups:
- Phase 2 Photobiomodulation (PBM): 670nm wavelength device twice a day for 90 seconds through 4 months. At the 4-month visit, participants who have not already received alternative treatments for DME will return the original device and receive the alternative treatment group device (i.e. the sham group will receive an active treatment device and the active treatment group will receive a sham device).
  Retilux: 670nm wavelength light
- Phase 2 Placebo: Broad spectrum light device twice a day for 90 seconds through 4 months. At the 4-month visit, participants who have not already received alternative treatments for DME will return the original device and receive the alternative treatment group device (i.e. the sham group will receive an active treatment device and the active treatment group will receive a sham device)
  Sham Light Device: Broad spectrum light device
Arm/Group | Phase 2 Photobiomodulation (PBM) | Phase 2 Placebo
Number analyzed (Participants) | 61 | 62
Number analyzed (Eyes) | 61 | 62
microns | -1 (44) | -2 (41)

ADVERSE EVENTS:
Time Frame: 8 Months
Groups:
- Phase 1 Photobiomodulation (PBM) Intervention: 670nm wavelength device twice a day for 90 seconds through 4 months. At the 4-month visit, participants who have not already received alternative treatments for DME will return the original device and receive the alternative treatment group device (i.e. the sham group will receive an active treatment device and the active treatment group will receive a sham device).
- Phase 1 Placebo Intervention: Broad spectrum light device twice a day for 90 seconds through 4 months. At the 4-month visit, participants who have not already received alternative treatments for DME will return the original device and receive the alternative treatment group device (i.e. the sham group will receive an active treatment device and the active treatment group will receive a sham device)
- Phase 2 Photobiomodulation (PBM) Intervention: 670nm wavelength device twice a day for 90 seconds 4 to 8 months. At the 4-month visit, participants who have not already received alternative treatments for DME will return the original device and receive the alternative treatment group device (i.e. the sham group will receive an active treatment device and the active treatment group will receive a sham device)
- Phase 2 Placebo Intervention: Broad spectrum light device twice a day for 90 seconds 4 to 8 months. At the 4-month visit, participants who have not already received alternative treatments for DME will return the original device and receive the alternative treatment group device (i.e. the sham group will receive an active treatment device and the active treatment group will receive a sham device)
Arm/Group | Phase 1 Photobiomodulation (PBM) Intervention | Phase 1 Placebo Intervention | Phase 2 Photobiomodulation (PBM) Intervention | Phase 2 Placebo Intervention
All-Cause Mortality (participants affected / at risk) | 1/69 | 0/66 | 0/61 | 2/62
Serious Adverse Events (participants affected / at risk) | 5/69 | 9/66 | 4/61 | 1/62
Other Adverse Events (participants affected / at risk) | 12/69 | 7/66 | 8/61 | 6/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Phase 1 Photobiomodulation (PBM) Intervention (N=69) | Phase 1 Placebo Intervention (N=66) | Phase 2 Photobiomodulation (PBM) Intervention (N=61) | Phase 2 Placebo Intervention (N=62)
Congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pressure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Water retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Broken bones (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fainting (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis of arm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stroke - Ischemic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.01% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Photobiomodulation (PBM) Intervention (N=69) | Phase 1 Placebo Intervention (N=66) | Phase 2 Photobiomodulation (PBM) Intervention (N=61) | Phase 2 Placebo Intervention (N=62)
Blepharitis (eyelid irritation) (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blepharo conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blurry vision (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Color vision change (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cotton wool spots (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic macular edema (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (3)
Eye ache (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye itching (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye tearing (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid margin crusting (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Macular edema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nuclear sclerosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Posterior vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensitivity to light (photophobia) (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Superficial punctate keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision decreased (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning sensation in face (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT03866473/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT03866473/SAP_001.pdf
  • Informed Consent Form (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT03866473/ICF_002.pdf